CLINICAL TRIAL: NCT00125307
Title: Tacrolimus for the Treatment of Systemic Lupus Erythematosus With Membranous Nephritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2004.229-T; CRE-2004.229-T
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2008-05

CONDITIONS: Lupus Nephritis; Lupus Erythematosus, Systemic
Keywords: SLE; glomerulonephritis; immunosuppressive therapy; type V (membranous) lupus nephritis
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic; Glomerulonephritis | interventions — Tacrolimus

INTERVENTIONS:
Drug: tacrolimus

SUMMARY:
The investigators study the efficacy and safety of tacrolimus in the treatment of membranous nephritis secondary to systemic lupus erythematosus.

DETAILED DESCRIPTION:
Glomerulonephritis is one of the major disease manifestations of systemic lupus erythematosus (SLE). The treatment of membranous (type V) lupus nephritis, a subset that carries a high morbidity, remains unsatisfactory. Recent studies suggest that immunosuppressive therapy targeted against the calcineurin pathway of T-helper cells, for example, tacrolimus, may be effective in the treatment of primary membranous nephropathy. The investigators plan to conduct an open-label single-arm study of the efficacy and safety of tacrolimus in the treatment of membranous nephropathy secondary to SLE. Twenty patients with biopsy-proven membranous nephropathy secondary to SLE will be recruited. They will be treated with oral prednisolone and tacrolimus for 6 months, followed by 6 months of maintenance steroids alone. Proteinuria, renal function, clinical and serologic lupus activity will be monitored. Complete remission is defined as 24-hour urinary protein excretion to less than 0.5 gm/day. This study will explore the potential role of tacrolimus in the treatment of membranous lupus nephritis, which is usually resistant to conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the revised American College of Rheumatology criteria for SLE
* Have biopsy-proven membranous nephropathy secondary to SLE
* Nephrotic syndrome with proteinuria (> 3 g/day) and serum albumin < 30 g/dl, with or without active urinary sediments despite steroid therapy (with or without cytotoxic agents)
* Age over 18 with informed consent
* Female patients of child-bearing age and male patients who agree to maintain effective birth control practice during the study

Exclusion Criteria:

* Patient with abnormal liver function tests
* Patient with hepatitis B surface antigen or who is hepatitis C antibody positive
* Patient who is diabetic
* Patient who is receiving non-steroidal anti-inflammatory drugs (NSAIDs) or other agents known to influence urinary protein excretion
* Patient is allergic or intolerant to macrolide antibiotics or tacrolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-01; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour urinary protein excretion

SECONDARY OUTCOMES:
Development of renal flare
Development of non-renal flare

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk-Chun Szeto, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, Hong Kong